CLINICAL TRIAL: NCT05592821
Title: Clinical and Radiographic Evaluation of Bone and Tissue Level Single Unit Implants: Two-piece Abutment Concept
Status: Completed | Type: Observational
Sponsor: Berceste Guler (Other)
Responsible Party: Sponsor-Investigator, Berceste Guler, Associate Professor, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Other Study IDs: 2020/09-06
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Bone Loss, Alveolar; Dental Implant Failed
Keywords: Soft tissue level implants; Bone level implants; Marginal bone loss; Two-piece abutment concept
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: soft tissue level implants: In this study, it was planned to use 20 implants of the same brand, with a single implant in the bilateral posterior regions in 10 patients. While the bone level implant is placed on one side of the patients, the tissue level implant will be used on the other side. The study will be designed as split-mouth. The type of implant to be placed in the regions will be decided according to the amount of keratinized gingival level above the alveolar crest level. Soft tissue level implants are in this group
  Interventions: Procedure: dental implant placement
- Control Group: bone level implants: In this study, it was planned to use 20 implants of the same brand, with a single implant in the bilateral posterior regions in 10 patients. While the bone level implant is placed on one side of the patients, the tissue level implant will be used on the other side. The study will be designed as split-mouth. The type of implant to be placed in the regions will be decided according to the amount of keratinized gingival level above the alveolar crest level. Bone level implants are in this group
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement — In both groups, dental implants of the same brand will be placed into the bone with the same protocol.

SUMMARY:
Dental implants have become one of the most common treatments used for the rehabilitation of lost teeth. The success rate of dental implant treatment is quite high. One of the criteria used for long-term implant success is the evaluation of radiographic marginal bone loss. Implants are used at the bone and tissue level in implant treatment. In this study, it was planned to use 20 implants of the same brand, with a single implant in the bilateral posterior regions in 10 patients.The study will be designed as split-mouth. The implant will be placed at the bone level with the same protocol in the two edentulous areas and the flap will be closed primarily. After 3 months, the substructure of the two-piece abutment concept system will be placed in a region during the healing head placement stage, and the bone level implant will be converted to the tissue level. A conventional healing cap will be placed in the other area. Periapical radiographs will be taken from the patients who participated in our study, as in all implant patients, during the pre-surgical planning phase and after implant placement. With the control periapical radiographs to be taken as a result of one-year follow-up, the marginal bone loss amount in the implants will be evaluated using soft-ware. Clinical measurements will be taken in all patients at the prosthetic loading session and 1 year after loading.

DETAILED DESCRIPTION:
Dental implants have become one of the most common treatments used for the rehabilitation of lost teeth. The success rate of dental implant treatment is quite high. One of the criteria used for long-term implant success is the evaluation of radiographic marginal bone loss. Implants are used at the bone and tissue level in implant treatment. The effects of bone and tissue level implants and peri-implant keratinized mucosa on marginal bone loss have been studied in the literature. In 2018, Vianna conducted research on 40 implants, 20 at the bone level and 20 at the tissue level, in split mouth design in 20 chronic periodontitis patients. Insufficient height of the peri-implant keratinized mucosa may cause sensitivity and pain during tooth brushing. This affects the patient's quality of life negatively, and also shortens the long-term survival of the implant as it may cause peri-implant alveolar bone loss and inflammation due to plaque deposition. It is known that the width of the keratinized gingiva decreases anatomically from anterior to posterior.

In this study, it was planned to use 20 implants of the same brand, with a single implant in the bilateral posterior regions in 10 patients.The study will be designed as split-mouth. The implant will be placed at the bone level with the same protocol in the two edentulous areas and the flap will be closed primarily. After 3 months, the substructure of the two-piece abutment concept system will be placed in a region during the healing head placement stage, and the bone level implant will be converted to the tissue level. A conventional healing cap will be placed in the other area. Before starting the surgery, after anesthesia is given, the width of the patient's peri-implant keratinized mucosa and the gingival height at the top of the alveolar crest will be measured. Periapical radiographs will be taken from the patients who participated in our study, as in all implant patients, during the pre-surgical planning phase and after implant placement. With the control periapical radiographs to be taken as a result of one-year follow-up, the marginal bone loss amount in the implants will be evaluated using soft-ware. Clinical measurements will be taken in all patients at the prosthetic loading session and 1 year after loading.

Clinical measurements

1. Plaque index (Löe & Silness) and gingival index (Silness & Löe) are obtained by measuring 4 regions of a tooth (mesial, distal, buccal and lingual) with a Williams periodontal probe.

   Attachment loss: It is the value of the distance between a tooth and the free gingiva, based on the enamel-cementum junction, measured using a Williams periodontal probe.
2. Bleeding on probing index (Ainamo & Bay): In this index, probing is performed by gently walking around the pocket. As a result of probing, the evaluation is made by looking at the presence or absence of bleeding in the gingiva. A positive value is given if bleeding occurs within 10-15 seconds after probing in the mesial, distal, buccal and lingual gingival parts of all teeth. The ratio of the bleeding area to the examined area is expressed as %.
3. Keratinized gingival width: It is the distance from the free gingival margin to the mucogingival junction line.
4. Vertical mucosal thickness: It is the distance from the apex of the alveolar crest to the gingival margin. It will be measured with a standardized William type probe.
5. Pocket depth: The vertical distance between the base of the periodontal sulcus and the gingival margin with a standard periodontal probe.
6. Peri-implant pocket depth: It is the vertical distance between the base of the peri-implant sulcus and the gingival margin.
7. Marginal bone level: Radiographic evaluation of the distance between the restoration margin and the bone level

Sample Selection: Taking the effect size of 0.08 for the significance value in the G Power analysis program as a reference to a previously presented study, 20 patients and 40 implants were planned to be taken for α= 0.05 and 80% power.

Statistical analysis method: All analyzes will be done with the (Statistical Package for the Social Sciences) SPSS software program. In-group temporal evaluations in test and control groups will be evaluated using Paired sample -T or Wilcoxon test according to normal distribution values. For comparisons between groups, the data will be analyzed with the Independent sample-T or Mann Whitney U test according to the normal distribution. The normal distribution of the data will be evaluated with the Kolmogorov-Smirnov test. Relationships between variables will be evaluated with Logistic Regression Analysis or Multivariate Regression Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* The patient does not have any systemic disease
* Implants are placed in the fully healed alveolar bone
* There is no need for horizontal and vertical augmentation in the area where the implant will be placed.
* Interocclusal distance greater than 7 mm
* The edentulous space is free-ended or the mesiodistal width in the interdental region is at least 6 mm
* Cooperative patients
* At least 9 mm of alveolar bone in the patient's mandible or maxilla in the area where the implant will be placed

Exclusion Criteria:

* Pregnant and breastfeeding women
* Mentally retarded patients
* Patients with immediate loading
* Patients with lesions in the alveolar bone
* Patients who smoke more than 10 cigarettes per day
* Patients who use drugs that suppress the immune system or impair recovery
* Patients using drugs that disrupt bone metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apply to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Peri-implant marginal bone loss. | 1 year following prosthetic restoration.
  Comparison of the 2 groups in terms of the amount of marginal bone loss.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler, Principal Investigator — Kütahya Health Sciences University Faculty of Dentistry
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) will be shared if the principal investigator is contacted.
Supporting Information: Study Protocol, CSR
Time Frame: After the research paper is published.
Access Criteria: The IPD will be shared if the principal investigator is contacted.

REFERENCES:
- [Result] Fernandez-Formoso N, Rilo B, Mora MJ, Martinez-Silva I, Diaz-Afonso AM. Radiographic evaluation of marginal bone maintenance around tissue level implant and bone level implant: a randomised controlled trial. A 1-year follow-up. J Oral Rehabil. 2012 Nov;39(11):830-7. doi: 10.1111/j.1365-2842.2012.02343.x. Epub 2012 Aug 13. PMID 22889084
- [Result] Lopez MA, Andreasi Bassi M, Confalone L, Gaudio RM, Lombardo L, Lauritano D. Retrospective study on bone-level and soft-tissue-level cylindrical implants. J Biol Regul Homeost Agents. 2016 Apr-Jun;30(2 Suppl 1):43-8. PMID 27469547
- [Derived] Ayyildiz BG, Terzioglu B, Bayindir BC. The Effect of Two-Piece Abutment Concept and Abutment Reconnection/Disconnection on Marginal Bone Level Changes: A Split-Mouth Randomized, Parallel-Designed, 36-Month Follow-Up, Preliminary Clinical Study. Int J Oral Maxillofac Implants. 2025 Sep 4;0(0):1-28. doi: 10.11607/jomi.11454. Online ahead of print. PMID 40907027